CLINICAL TRIAL: NCT06656078
Title: The Effects of Different Types of Cognitive Load on Gait
Brief Title: Comparison of Effect of Different Methods of Cognitive Loading on Gait of Normal Healthy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: REC/01885 Imran Amjad
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Load, Performance

STUDY DESIGN:
Intervention Model Description: Research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 male (Experimental): All members of group number 1 who fall in the eligibility criteria will undergo three different types of cognitive loading.
  Three types of cognitive loading will be applied randomly to eliminate any bias.
  Each Method will be applied three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. WORKING MEMORY TASK:; Other: 2. VISUAL AND VERBAL FLUENCY TASK; Other: 3. MOTOR TASK:
- Group 2 female (Experimental): All members of group number 2 who fall in the eligibility criteria will undergo three different types of cognitive loading.
  Three types of cognitive loading will be applied randomly to eliminate any bias.
  Each Method will be applied three times along with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. WORKING MEMORY TASK:; Other: 2. VISUAL AND VERBAL FLUENCY TASK; Other: 3. MOTOR TASK:

INTERVENTIONS:
Other: 1. WORKING MEMORY TASK: — Arithmetic task: backward counting with serial 3 subtractions out loud. Group 1 and Group 2 participants will be asked to count backwards with serial 3 subtractions out loud while walking 10 meters. There is considerable disruption of performance because of simultaneous articulatory suppression. However, when errors were observed they were calculated to be numerically close to the correct figure which suggests that performance was not completely disrupted by suppression of articulation.
Other: 2. VISUAL AND VERBAL FLUENCY TASK — Modified Stroop test or Stroop colour word test: Participants are asked to name the colour of ink that each word is printed. It is the most frequent test used to show attention bias in anxiety patients. This test will appear on the mobile phone in their hands while they walk to increase the effect of cognitive loading.
Other: 3. MOTOR TASK: — Carrying a tray with four glasses filled with water. Participants will be asked to hold a tray of glasses filled with water and walk 10 meters to calculate the effect of cognitive loading on gait.

SUMMARY:
Comparison of effect of different methods of cognitive loading on gait of normal healthy students.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students from colleges of Abbottabad.
* Age limit (17 to 20) According to (FSC admission criteria age of the student should not be more than 18 to enter the college.)
* Healthy individuals without any neurological and MSK disorder. (screening will be done before performing the test on the student, questions regarding the above-mentioned conditions and consent will be signed before starting the test)

Exclusion Criteria:

* Any student with visible physical deformity or MSK disorder will not be included in this research (15)
* Any student with a psychiatric or neurological disorder will not be included (16)
* Any student with cardiac abnormality will be excluded from this research (17)
* Any student who does not fall in this age group will not be included in this research.
* Colleges outside Abbottabad will not be included in this research.

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All male and female healthy students are eligible to participate.
Enrollment: 82 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Walking speed (m/s) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures the walking speed with moderate to excellent reliability while the participant is walking normally with (ICC=0.93). Walking speed usually decreases if the participant performs a task that challenges dynamic balance.
Walking speed (m/s) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures the walking speed with moderate to excellent reliability while the participant is walking normally with (ICC=0.93). Walking speed usually decreases if the participant performs a task that challenges dynamic balance.
Walking speed (m/s) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures the walking speed with moderate to excellent reliability while the participant is walking normally with (ICC=0.93). Walking speed usually decreases if the participant performs a task that challenges dynamic balance.
Gait symmetry (%) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures gait symmetry with moderate to excellent reliability while the participant is walking normally with (ICC=0.65) Gait symmetry tends to decrease if the participant undergoes a task that includes dynamic balance.
Gait symmetry (%) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures gait symmetry with moderate to excellent reliability while the participant is walking normally with (ICC=0.65) Gait symmetry tends to decrease if the participant undergoes a task that includes dynamic balance.
Gait symmetry (%) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures gait symmetry with moderate to excellent reliability while the participant is walking normally with (ICC=0.65) Gait symmetry tends to decrease if the participant undergoes a task that includes dynamic balance.
Step length(m) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures step length with moderate to excellent reliability while the participant is walking normally with (ICC=0.94). Step length usually increases with challenged dynamic balance-based activities.
Step length(m) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step length with moderate to excellent reliability while the participant is walking normally with (ICC=0.94). Step length usually increases with challenged dynamic balance-based activities.
Step length(m) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step length with moderate to excellent reliability while the participant is walking normally with (ICC=0.94). Step length usually increases with challenged dynamic balance-based activities.
Step time(s) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to excellent reliability while the participant is walking normally with (ICC=0.84). Step time increases under the effect of dynamic balance-based activities.
Step time(s) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to excellent reliability while the participant is walking normally with (ICC=0.84). Step time increases under the effect of dynamic balance-based activities.
Step time(s) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to excellent reliability while the participant is walking normally with (ICC=0.84). Step time increases under the effect of dynamic balance-based activities.
Step time variability(%) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to poor reliability while the participant is walking normally (ICC=0.51). Step time variability tends to increase if a participant undergoes dynamic balance-based activities.
Step time variability(%) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to poor reliability while the participant is walking normally (ICC=0.51). Step time variability tends to increase if a participant undergoes dynamic balance-based activities.
Step time variability(%) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time with moderate to poor reliability while the participant is walking normally (ICC=0.51). Step time variability tends to increase if a participant undergoes dynamic balance-based activities.
Step length variability(%) | Baseline
  For gait activity, the G&B app measures step length variability with moderate to poor reliability while the participant is walking normally (ICC=0.16). step length variability tends to increase with activities that involve dynamic balance.
Step length asymmetry(%) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step length asymmetry with moderate to poor reliability while the participant is walking normally with (ICC=0.6). Step length asymmetry tends to increase with tasks that include dynamic balance.
Step length asymmetry(%) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step length asymmetry with moderate to poor reliability while the participant is walking normally with (ICC=0.6). Step length asymmetry tends to increase with tasks that include dynamic balance.
Step time asymmetry(%) | Baseline
  For gait activity, the Gait and Balance mobile app (G&B) measures step time asymmetry with moderate reliability while the participant is walking normally with (ICC=0.68). Step time asymmetry tends to increase with activities that include dynamic balance.
Step time asymmetry(%) | During Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time asymmetry with moderate reliability while the participant is walking normally with (ICC=0.68). Step time asymmetry tends to increase with activities that include dynamic balance.
Step time asymmetry(%) | Immediately after Cognitive loading tests
  For gait activity, the Gait and Balance mobile app (G&B) measures step time asymmetry with moderate reliability while the participant is walking normally with (ICC=0.68). Step time asymmetry tends to increase with activities that include dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No